CLINICAL TRIAL: NCT01146964
Title: Comparison of Manual Super Small Incision Cataract Surgery and Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangtian Zhou, MD, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10003
Record Dates: First submitted 2010-06-02; First posted 2010-06-22 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Cataract; Phacoemulsification
Keywords: Age related cataract; Phacoemulsification; Manual super small incision cataract surgery
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phacoemulsification, Safety, Efficacy (Experimental)
  Interventions: Procedure: Phacoemulsification
- MSSICS, Safety, Efficacy (Experimental)
  Interventions: Procedure: MSSICS

INTERVENTIONS:
Procedure: MSSICS — Manual super small incision cataract surgery
  Arms: MSSICS, Safety, Efficacy
Procedure: Phacoemulsification — cataract surgery with Phacoemulsification
  Arms: Phacoemulsification, Safety, Efficacy

SUMMARY:
The purpose of this study is to compare the safety and efficacy of manual super small incision cataract surgery (MSSICS) and Phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* Age related cataract patients
* Cataract density grade II-III according to the Emery-Little system classification system

Exclusion Criteria:

* Legal guardian(s) is/are not present for permission
* Other eye diseases impairing visual acuity (ie. glaucoma)
* patients with severe systemic diseases not good for ocular surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Corneal endothelial cell loss | 3 months postoperatively

SECONDARY OUTCOMES:
postoperative astigmatism | 3 months postoperatively
visual acuity | 3 month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, MD, PhD, Principal Investigator — Eye Hospital, Wenzhou Medical College, China
Locations (1):
- Eye Hospital, Wenzhou Medical College, Wenzhou, Zhejiang, China